CLINICAL TRIAL: NCT06191380
Title: Effects of a Single Bout of Moderate Intensity Aerobic Cycling Exercise Combined With Virtual Reality on Processing Speed in Persons With Multiple Sclerosis and Mobility Disability
Brief Title: Effects of Cycling and Virtual Reality on Thinking Speed in Persons With MS (PACE-MS)
Acronym: PACE-MS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kessler Foundation (Other)
Collaborators: Consortium of Multiple Sclerosis Centers (Other)
Responsible Party: Principal Investigator, Carly Wender, Research Scientist, Kessler Foundation
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: R123723
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Leg Cycling; Virtual Reality; Mobility Disability; Processing Speed
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Masking Description: Participants will be blinded to the hypothesized effect of each exercise condition.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cycling Alone (Active Comparator): Cycling alone, with no virtual reality.
  Interventions: Behavioral: PACE-MS
- Cycling with Visually Stimulating VR (Experimental): Cycling with virtual reality where I only have to look at the environment while I cycle.
  Interventions: Behavioral: PACE-MS
- Cycling with Cognitively Stimulating VR (Experimental): Cycling with virtual reality where I have to complete a thinking task while cycling in the virtual environment.
  Interventions: Behavioral: PACE-MS

INTERVENTIONS:
Behavioral: PACE-MS — A single bout of cycling.

SUMMARY:
To compare the effects of cycling exercise with different types of virtual reality on processing/thinking speed in persons with multiple sclerosis (MS).

DETAILED DESCRIPTION:
The purpose of this research study is to learn how different types of cycling exercise can improve short-term processing speed, or speed of thinking, in persons with MS. In this study, we will compare the effects of cycling alone to cycling with two different types of virtual reality. Participants will complete all three cycling conditions, one per week. We are studying these types of cycling because there are currently no effective treatment options to improve processing speed in persons with MS and combining exercise with virtual reality is a promising technique.

ELIGIBILITY:
Inclusion Criteria:

* Speak English as their primary language
* Confirmed MS diagnosis by a neurologist
* Be relapse and steroid-free for at least 30 days
* Mild-to-moderate self-report mobility disability

Exclusion Criteria:

* History of neurological disorders besides MS or history of uncontrolled psychiatric disorders (ex: major depression)
* Have contraindications to exercise, based on the Physical Activity Readiness Questionnaire (PAR-Q)
* Currently use medications that may impact cognition (ex: steroids, benzodiazepines)
* Currently pregnant
* Severe cognitive impairment as measured by the Modified Telephone Interview of Cognitive Status (TICS-M)
* No indication of age-related mild cognitive impairment or dementia, based on the MOCA-Blind (i.e., MOCA-Blind ≥19).
* High likelihood of motion sickness
* Regular cyclist, defined as cycling for at least 150 minutes/week

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2024-02-12 (Actual); Primary Completion 2025-10-28 (Actual); Study Completion 2025-10-28 (Actual)

PRIMARY OUTCOMES:
Modified Flanker Task (MFT) | Immediately before the single bout of cycling and 5 minutes after the single bout of cycling.
  Response time on a computerized test is conceptualized as a measure of processing speed. Participants are tasked with identifying the direction of the central target stimulus that is flanked by either congruent (<<<<<) or incongruent (>><>>) stimuli by pressing the correct keyboard key.

SECONDARY OUTCOMES:
Baseline mobility disability | Baseline visit only
  Mobility disability status will be measured with a neurological exam to get an EDSS score.
Baseline Symbol Digit Modalities Test (SDMT) | Baseline visit only.
  Processing speed will be measured with the SDMT as a more stable measure of processing speed.

CONTACTS AND LOCATIONS:
Overall Officials: Carly Wender, PhD, Principal Investigator — Kessler Foundation
Locations (1):
- Kessler Foundation, East Hanover, New Jersey, United States

IPD SHARING:
Plan to Share IPD: Undecided